CLINICAL TRIAL: NCT05572905
Title: Novel Approaches to Enhance Insulin-sensitizing Effects of Exercise: Targeting PAHSA Metabolism
Brief Title: Effect of Acute Bout of Exercise on Levels of PAHSA
Acronym: ETAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lenka Rossmeislova (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); Czech Academy of Sciences (Other)
Responsible Party: Sponsor-Investigator, Lenka Rossmeislova, Principal Investigator, Head of Laboratory of Physiology and Pathophysiology of Adipose Tissue, Department of Pathophysiology, Third Faculty of Medicine, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NU21-01-00469
Record Dates: First submitted 2022-09-26; First posted 2022-10-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Insulin Sensitivity
Keywords: acute exercise; adipose tissue; insulin sensitivity; PAHSA; lipokines; FAHFA
MeSH Terms: conditions — Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single groups assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young lean men and women (Experimental): 25 to 40 y.o. participants with body mass index in range of 18.5 to 25
  Interventions: Other: Exercise; Other: Fasting control
- Young obese men and women (Experimental): 25 to 40 y.o. participants with body mass index in range of 30 to 45.
  Interventions: Other: Exercise; Other: Fasting control
- Elderly men and women (Experimental): 65 to 80 y.o. participants with body mass index in range of 18.5 to 30.
  Interventions: Other: Exercise; Other: Fasting control

INTERVENTIONS:
Other: Exercise — Patients after overnight fast will cycle on ergo-meter for 60 minutes. No per-oral food intake will be allowed during the test. Level of the intensity of exercise will be determined as individual range of heart frequency (HF), oxygen consumption (VO2) and respiratory quotient (RQ) just bellow the aerobic threshold of the given participant (close to anticipated fatmax). These values will be obtained during maximal capacity stress test on cyclo-ergo-meter. This maximum stress test will be performed at least one week prior to the 60 minutes exercise to eliminate potential carry-over effect. Power output will be modulated during the 60 minutes of exercise to ensure keeping participants values of HF, RQ and VO2 in the given range. Blood will be sampled at 5 time points with interval of 30 minutes during the exercise (0, 30, 60, 90, 120) and 24 hours post-exercise.
Other: Fasting control — The same participants will be monitored while resting for 120 minutes in calm environment. No peroral food intake will be allowed during the test. Fasting control will take place at least one week apart of the exercise. Blood will be sampled at 5 timepoints with interval of 30 minutes during the exercise (0, 30, 60, 90, 120) and 24 hours post-control.

SUMMARY:
Exercise represents an important tool in the prevention and treatment of metabolic disorders associated with obesity and aging, such as type 2 diabetes and cardiovascular disease. Besides skeletal muscle and its myokinins, the metabolic effects of exercise also rely on the induction of favorable changes in adipose tissue function. For example, adipose tissue is a source of lipokinins from the family of palmitic acid esters of hydroxy fatty acids (PAHSA), which have anti-inflammatory and insulin-sensitizing properties. We have recently shown that 4 months of exercise training increases PAHSA levels in adipose tissue and circulation. However, the mechanisms involved in the induction of PAHSA levels in response to exercise are unknown. The aim of the Effect of Acute Bout of Exercise on Levels of PAHSA (ETAPA) project is therefore to investigate the regulation of PAHSA metabolism in response to both acute and chronic exercise. To achieve this goal, we will employ state-of-the-art analytical methods to measure PAHSA levels in both adipose tissue and circulation of subjects of various ages and adiposity status. The main output of the ETAPA project will be the proof of principle regarding the important role of PAHSA lipokinins in exercise-induced enhancement of insulin sensitivity and the identification of potential drug targets that could be used to further improve PAHSA metabolism for the treatment of metabolic disorders associated with aging or obesity.

ELIGIBILITY:
Inclusion Criteria:

* healthy young lean, young obese and older omnivorous men and women as defined by BMI, self-reported activity, self-reported medical history and self-reported diet assessment
* must be able to withstand repeated blood draws
* must be able to undergo abdominal fat biopsy

Exclusion Criteria:

* use of betablockers
* use of glucocorticoids
* use of non-steroidal anti-inflammatory drugs
* use of metformin in prediabetes
* use of psychiatric drugs such as selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors, anticonvulsants and others
* oncologic malignancy
* chronic inflammatory or autoimmune diseases
* diabetes mellitus
* chronic ischemic heart disease
* cardiovascular and pulmonary disease
* renal and hepatological disease as assessed per biochemistry
* musculo-skeletal deviations limiting physical performance
* substance abuse
* other than omnivorous diet

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Assessment of PAHSA levels and its changes in response to exercise and fasting in cohorts differing in age and fat mass | 2 years
  PAHSA levels [nmol/l] in serum sampled at pre-set time-points during control and intervention visits (including exercise session or plain fasting) and in subcutaneous abdominal white adipose tissue will be assessed by quantitative targeted lipidomic analysis.
  Absolute and fold-change of PAHSA in plasma induced by experimental intervention (exercise, fasting) will be compared among individual cohorts.

SECONDARY OUTCOMES:
Correlation of PAHSA levels with anthropometry and clinical characteristics | 2 years
  Basal levels of PAHSA and its changes in response to interventions will be correlated with anthropometric parameters (age, weight, fat mass) and parameters of physical fitness. Fat mass will be assessed by dual energy X-ray absorptiometry. Intercohort matching of obese and elderly subjects based on fat mass will be improved throughout the recruitment phase by utilization of fat mass assessment on two distinct certified bioimpedance instruments. Cohort physical fitness will be calculated as average from individual VO2max values obtained from maximum ergometry testing. Intercohort matching of young lean and young obese men and women will be based on age.
Correlation of PAHSA with various indexes of insulin sensitivity | 2 years
  Basal levels of PAHSA and its changes in response to interventions will be correlated with indices of muscle insulin sensitivity (MISI), hepatic insulin resistance (HIRI), adipose tissue insulin resistance (Adipo-IR) and homeostatic model assessment of insulin resistance (HOMA-IR). Values for measurement will be obtained by biochemical analysis of blood sampled during 5-point oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Lenka Rossmeislová, PhD, Principal Investigator — 3rd Faculty of Medicine of Charles University in Prague
Locations (1):
- 3rd faculty of medicine, Charles University, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brezinova M, Kuda O, Hansikova J, Rombaldova M, Balas L, Bardova K, Durand T, Rossmeisl M, Cerna M, Stranak Z, Kopecky J. Levels of palmitic acid ester of hydroxystearic acid (PAHSA) are reduced in the breast milk of obese mothers. Biochim Biophys Acta Mol Cell Biol Lipids. 2018 Feb;1863(2):126-131. doi: 10.1016/j.bbalip.2017.11.004. Epub 2017 Nov 14. PMID 29154942
- [Result] Paluchova V, Oseeva M, Brezinova M, Cajka T, Bardova K, Adamcova K, Zacek P, Brejchova K, Balas L, Chodounska H, Kudova E, Schreiber R, Zechner R, Durand T, Rossmeisl M, Abumrad NA, Kopecky J, Kuda O. Lipokine 5-PAHSA Is Regulated by Adipose Triglyceride Lipase and Primes Adipocytes for De Novo Lipogenesis in Mice. Diabetes. 2020 Mar;69(3):300-312. doi: 10.2337/db19-0494. Epub 2019 Dec 5. PMID 31806624
- See also: Related Info — https://www.lf3.cuni.cz/3LF-108.html?news=17665&locale=cz